CLINICAL TRIAL: NCT01440660
Title: Phenotypes of Nonproliferative Diabetic Retinopathy in Diabetes Type 2 Patients Identified by Optical Coherence Tomography, Colour Fundus Photography, Fluorescein Leakage and Multifocal Electrophysiology (DIAMARKER Project: Genetic Susceptibility for Multi-systemic Complications in Diabetes Type-2: New Biomarkers for Diagnostic and Therapeutic Monitoring).
Brief Title: Phenotypes of Nonproliferative Diabetic Retinopathy in DM 2 Patients Identified by OCT, CFP, RLA and mfERG (DIAMARKER)
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: University of Coimbra (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2011-01
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Type-2 Diabetes; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Leaking Phenotype: Retinal thickness (RT) increase (increase in RT above normal range as measured by OCT, considering the macular thickness normative data) in the central subfield, the inner ring and/or the outer ring.
- Ischemic Phenotype: Neovascular disease activity as shown by microaneurysms (MA) turnover (MA formation rate >= 2, i.e. number of new MA per year) computed from CFP using the RetmarkerDR software.

SUMMARY:
To characterise phenotypes of Non Proliferative Diabetic Retinopathy (NPDR) progression using multimodal testing/imaging procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years-old.
2. Diabetes mellitus type 2 according to 1985 WHO criteria.
3. Non-proliferative diabetic retinopathy (ETDRS level <= 35)
4. Signs of NPDR progression based on existing clinical information:

   1. Retinal thickness (RT) increase (increase in RT above normal range as measured by OCT, considering the macular thickness normative data) in the central subfield, the inner ring and/or the outer ring (leaking phenotype); OR
   2. Neovascular disease activity as shown by microaneurysms (MA) turnover (MA formation rate >= 2, i.e. number of new MA per year) computed from CFP using the RetmarkerDR software (ischemic phenotype).
5. Informed consent.

Exclusion Criteria:

1. Cataract or other eye disease that may interfere with fundus examinations
2. Any eye surgery or treatment within a period of 6-months.
3. Pregnant or nursing (lactating) women.
4. Patients with chronic or severe kidney disease (glomerular filtration rate, GFR < 30 mL/min/1.73m2).
5. Patients with acute kidney injury.
6. Patients with known allergic or hypersensitivity reactions to gadolinium, versetamide or any of the inert ingredients.
7. Patients around the time of liver transplantation..
8. Patients with implants containing metals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 20 patients, male and female over 18 years-old, with type-2 diabetes mellitus and NPDR with signs of DR progression (RT increase and/or MA turnover) (according to the inclusion/exclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Multimodal testing/imaging procedures - Ophthalmological Imaging | 24 months
  Retinal thickness measured with OCT;
Multimodal testing/imaging procedures - Ophthalmological Imaging | 24 months
  MA turnover computed based on CFP.
Multimodal testing/imaging procedures - Ophthalmological Imaging | 12 months
  Macular area with increased retinal fluorescein leakage based on RLA.
Multimodal testing/imaging procedures - Ophthalmological Imaging | 12 months
  Implicit time local and ring amplitudes measured with mfERG.
Multimodal testing/imaging procedures - Psychophysical Testing | 12 months
  Psychophysical tests for speed discrimination, achromatic contrast, and chromatic contrast.
Multimodal testing/imaging procedures - Barin Imaging | 12 months
  Perfusion change measured with ASL.
Multimodal testing/imaging procedures - Ophthalmological Imaging | 12 months
  Blood-Brain Barrier alterations assessed contrast agent with Dynamic MR.
Multimodal testing/imaging procedures - Brain Imaging | 12 months
  Metabolite concentrations assessed with MR Spectroscopy.

SECONDARY OUTCOMES:
Multimodal testing/ imaging modalities (raw data) | 24 months
  Raw data obtained from the different modalities (OCT,MA turnover, RLA,mfERG, psychophysical tests, ASL, Dynamic MR and MR Spectroscopy).

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD PhD, Study Chair — Association for Innovation and Biomedical Research on Light and Image; Miguel Castelo-Branco, MD PhD, Study Chair — FMUC; Luísa Ribeiro, MD MSc, Principal Investigator — AIBILI - CEC
Locations (1):
- AIBILI - Clinical Trials Centre (CEC), Coimbra, Portugal